CLINICAL TRIAL: NCT04115384
Title: A Single Center Feasibility Study of Intranasal Insulin in Frontotemporal Dementia NIFT-D
Brief Title: Intranasal Insulin in Frontotemporal Dementia (FTD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID - unable to restart after restrictions were lifted
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A18-305
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Results first posted 2023-07-06 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-04

CONDITIONS: Frontotemporal Dementia, Behavioral Variant
Keywords: intranasal; insulin
MeSH Terms: conditions — Pick Disease of the Brain; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Insulin (Novolin-R) (Experimental): Regular insulin (Novolin-R) 20 IU/IN (0.1ml/10 units IN in each nostril) BID
  Interventions: Drug: Novolin-R insulin

INTERVENTIONS:
Drug: Novolin-R insulin — Insulin (Novolin-R) 20 IU/IN (0.1ml/10 units IN in each nostril), twice per day, once in the morning and again in the evening (at least 8 hours between doses) for 4 weeks.
  Other Names: insulin, Novolin-R

SUMMARY:
This project will study intranasal (IN) insulin in Frontotemporal dementia (FTD) in 12 patients. Study Investigators aim to evaluate the feasibility of the EXAMINER cognitive battery as a cognitive outcome measure in FTD, the ability of the HealthPartners Center for Memory and Aging's ability to sufficiently recruit subjects with FTD, and the safety of IN regular insulin administered 20 IU twice per day in two specific variants of FTD (behavioral variant frontotemporal dementia (bv-FTD), semantic dementia (SD)) over a 4 week period.

DETAILED DESCRIPTION:
Frontotemporal dementia (FTD) with its multiple pathological manifestations, is a disease that results in progressive deterioration of social comportment, executive function, and language. Despite the debilitating nature of FTD and the relatively high prevalence in the younger patient population, available pharmacological interventions are limited to symptomatic treatments. There are no therapeutic agents that have been developed that specifically treat the progressive cognitive symptoms of FTD. This project will study IN insulin in FTD in 12 patients. Investigators aim to evaluate the feasibility of the EXAMINER cognitive battery as a cognitive outcome measure in FTD, the ability of the HealthPartners Center for Memory and Aging's Center's ability to sufficiently recruit subjects with FTD, and the safety of IN regular insulin administered 20 IU twice per day in two specific variants of FTD (behavioral variant frontotemporal dementia (bv-FTD), semantic dementia (SD)) over a 4 week period. Frontotemporal dementia (FTD) with its multiple pathological manifestations, is a disease that results in progressive deterioration of social comportment, executive function, and language. Despite the debilitating nature of FTD and the relatively high prevalence in the younger patient population, available pharmacological interventions are limited to symptomatic treatments. There are no therapeutic agents that have been developed that specifically treat the progressive cognitive symptoms of FTD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject meeting international consensus criteria for probable behavioral variant frontotemporal dementia or criteria for semantic dementia (Gorno-Tempini et al., 2011; Rascovsky et al., 2011)
2. Subject has a Mini-Mental State Exam (MMSE) score ≥18.
3. Subject is > 40 and <90 years of age.
4. Female subjects are post-menopausal or have a negative pregnancy test
5. The subject must be proficient in speaking, reading and understanding English in order to comply with procedural testing of cognitive function, memory and physiology.
6. Subject has a dedicated family member/caregiver, who will be able to attend all visits and report on subject's status.
7. Subject and family member/caregiver have both provided fully informed written consent prior to participation. In the event that subject is legally unable to provide informed written consent due to deterioration in cognitive abilities, fully informed written consent must be provided by a legally authorized representative.
8. Subject must have undergone a brain computed tomography (CT) scan or magnetic resonance imaging (MRI) scan as part of receiving frontotemporal dementia (FTD) diagnosis

Exclusion Criteria:

1. Subject has medical history and/or clinically determined evidence of other central nervous system (CNS) disorders including, but not limited to brain tumor, active subdural hematoma, seizure disorder, multiple sclerosis, Alzheimer's disease, vascular dementia, corticobasal syndrome, progressive supranuclear palsy, Parkinson's disease, multiple system atrophy, Lewy body dementia, normal pressure hydrocephalus, Huntington's disease, or Jakob-Creutzfeldt disease presenting as dementia.
2. Subject has medical history and/or clinically determined disorders: current B12 deficiency, chronic sinusitis, untreated thyroid disease, or significant head trauma.
3. Subject has history of any of the following: moderate to severe pulmonary disease, poorly controlled congestive heart failure, significant cardiovascular and/or cerebrovascular events within previous 6 months, condition known to affect absorption, distribution, metabolism, or excretion of drugs such as any hepatic, renal or gastrointestinal disease or any other clinically relevant abnormality that inclusion would pose a safety risk to the subject as determined by investigator.
4. Subject has had previous nasal and/or oto-pharyngeal surgery and severe deviated septum and/or other anomalies.
5. Subject has a history of any psychiatric illness that would pose a safety risk to the subject as determined by investigator.
6. Subject is currently taking any medications (anticholinergics, antihistamines, benzodiazepines, barbiturates, or insulin) that are clinically contraindicated as determined by investigator.
7. Subject has undergone a recent change (<1 month) in their selective serotonin reuptake inhibitors (SSRI) or anti-depressant medication.
8. Subject has current or recent drug or alcohol abuse or dependence as defined by the Diagnostic and Statistical Manual of Mental Disorders 5, Text Revision (DSM-IV TR).
9. Screening laboratory results that are medically relevant, in which inclusion would pose a safety risk to the subject as determined by investigator.
10. The subject has participated in a clinical trial investigation within 1 month of this study.
11. The subject has an insulin allergy.

Ages: 41 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Rosenbloom, MD, Principal Investigator — HealthPartners Neurology
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Insulin (Novolin-R)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Measured by EXAMINER Battery
Description: Number of patients completing the entire EXAMINER battery. Range: 0-3. More participants completing EXAMINER indicates higher feasibility.
Time Frame: Baseline and Post Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 3
Participants | 3

2. Primary Outcome: Feasibility Measured by Recruitment
Description: Number of patients enrolled in this study. Range: 0-12. More participants enrolling indicates higher feasibility.
Time Frame: Baseline
Population: The original goal was to include 12 participants. Since this is a feasibility outcome, the analysis population is the original goal total.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 12
Participants | 3

3. Primary Outcome: Safety Measured by Total Serious Adverse Events (SAEs) and Adverse Events (AEs)
Description: Total number of AEs/SAEs during the course of treatment. More AEs/SAEs indicates a less safe treatment.
Time Frame: 2 months
Measure: Number; unit: Total number of AEs/SAEs reported
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 3
Total number of AEs/SAEs reported | 1

4. Secondary Outcome: Feasibility Measured by Completion of Study
Description: Number of patients completing the entire study. Range: 0-12. More participants completing the study indicates higher feasibility.
Time Frame: 2 months
Population: 12 participants were expected. Only 3 participants were able to complete the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 12
Participants | 3

5. Secondary Outcome: Feasibility Measured by Screen Fails
Description: Number of patients screen failing during the study. More participants screen failing the study indicates lower feasibility.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 3
Participants | 0

6. Secondary Outcome: Safety Measured by Unique Subjects With Serious Adverse Events (SAEs) and Adverse Events (AEs)
Description: Total number of unique participants experiencing AEs/SAEs during the course of treatment. More unique participants experiencing AEs/SAEs indicates a less safe treatment.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 3
Participants | 1

7. Other Pre Specified Outcome: Pre to Post Working Memory Measured by EXAMINER - Dot Counting
Description: Dot counting measures verbal working memory. Participants are asked to count colored shapes on a tables and remember the final total over 6 trials. Scores are totaled as the number of correct answers or the number of answers recalled. Range: 0-27. A higher score indicates better performance.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 3
score on a scale | 6.33 (3.06)

8. Other Pre Specified Outcome: Pre to Post Verbal Fluency Measured by EXAMINER - Animal Fluency
Description: Participants are asked to name as many animals as he/she can in 60 seconds. Scores are totaled as the number of animals verbalized. A higher score indicates better performance.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: named animals
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 3
named animals | -0.33 (3.21)

9. Other Pre Specified Outcome: Pre to Post Inhibition by EXAMINER - Flanker
Description: Participants are asked to choose the direction of one the center arrow in a group 5 arrows. Range: 0- 10. This is a global score that combines accuracy and reaction time. A higher score indicates better performance.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 3
score on a scale | -0.145 (0.26)

10. Other Pre Specified Outcome: Pre to Post Inhibition by EXAMINER - Set Shifting
Description: Participants are asked to match stimulus on different parts of a tablet screen. Range: 0- 10. This is a global score that combines accuracy and reaction time. A higher score indicates better performance.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: change is score on a scale
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 3
change is score on a scale | -0.36 (0.13)

11. Other Pre Specified Outcome: Pre to Post Appetite Changes by the Appetite and Eating Habit Questionnaire (APEHQ) - Swallowing Subscore
Description: A survey about changes in eating behaviors. The sum of frequency times severity of swallowing related questions is the score for this portion. Caregivers of participant are asked to fill this survey out. Range: 0-96. Higher scores indicate higher difficulty swallowing that produces conflict or embarrassment.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 3
change in score on a scale | 0.67 (0.53)

12. Other Pre Specified Outcome: Pre to Post Appetite Changes by the Appetite and Eating Habit Questionnaire (APEHQ) - Appetite Subscore
Description: A survey about changes in eating behaviors. The sum of frequency times severity of appetite related questions is the score for this portion. Caregivers of participant are asked to fill this survey out Range: 0-96. Higher scores indicate a greater change in appetite that produces conflict or embarrassment.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 3
change in score on a scale | -0.67 (1.53)

13. Other Pre Specified Outcome: Pre to Post Appetite Changes by the Appetite and Eating Habit Questionnaire (APEHQ) - Eating Habits Subscore
Description: A survey about changes in eating behaviors. The sum of frequency times severity of eating habit related questions is the score for this portion. Caregivers of participant are asked to fill this survey out Range: 0-72. Higher scores indicate a greater change in eating habits that produces conflict or embarrassment.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 3
change in score on a scale | 7 (11.3)

14. Other Pre Specified Outcome: Pre to Post Appetite Changes by the Appetite and Eating Habit Questionnaire (APEHQ) - Food Preference Subscore
Description: A survey about changes in eating behaviors. The sum of frequency times severity of food preference related questions is the score for this portion. Caregivers of participant are asked to fill this survey out Range: 0-84. Higher scores indicate a greater change in food preferences that produces conflict or embarrassment.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 3
change in score on a scale | 2.67 (4.62)

15. Other Pre Specified Outcome: Pre to Post Appetite Changes by the Appetite and Eating Habit Questionnaire (APEHQ) - Other Oral Behaviors Subscore
Description: A survey about changes in eating behaviors. The sum of frequency times severity of other oral behavior related questions is the score for this portion. Caregivers of participant are asked to fill this survey out Range: 0-60. Higher scores indicate a greater changes that produces conflict or embarrassment.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Insulin (Novolin-R)
Number analyzed (Participants) | 3
change in score on a scale | 0.33 (3.51)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Insulin (Novolin-R)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin (Novolin-R) (N=3)
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Persistent coughing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT04115384/Prot_SAP_000.pdf